CLINICAL TRIAL: NCT02079259
Title: CVP-guided Aquapheresis for the Treatment of Acute Congestion in Heart Failure - A Pilot Study to Optimize Individualized Volume Depletion
Brief Title: CVP-guided Aquapheresis for the Treatment of Acute Congestion in Heart Failure
Acronym: Aquadex
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Other Study IDs: Aquadex
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ultrafiltration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ultrafiltration

SUMMARY:
The number of patients with acute congestion on chronic heart failure is increasing. Ultrafiltration has recently been proposed as an alternative approach for the stabilization of volume balance, especially in patients with imminent diuretic resistance.

There is increasing evidence that ultrafiltration may relief cardiac congestion with lesser effects on blood pressure and activation of renin angiotensin system, respectively . However, recent studies revealed conflicting results: demonstration the superiority of ultrafiltration in comparison to diuretic treatment, and a lack of evidence of benefit, as well as an excess of adverse events with ultrafiltration.

Aquapheresis with adapted ultrafiltration rate guided by central venous pressure is safer than aquaphesis with a constant ultrafiltration with comparable effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure scheduled for LVAD
* Indication for CVVH/Aquapheresis

Exclusion Criteria:

* Renal Disease (GFR <20 ml / min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic heart failure listed for LVAD
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Changes in central venous pressure | Changes from Baseline to 48 h after intervention

SECONDARY OUTCOMES:
amount of net fluid loss | 48 h
Measure of dyspnea using a visual analog scale | Changes from Baseline to 48 h after intervention
heart function | 7 days
  right/left heart function measured by Echocardiography and BNP (Brain Natriuretic Peptide)
Biomarker | Changes from Baseline to 48 h after intervention
  GFR, Cystatin C, HCO3-, NT-proBNP, CK, Troponin, Hematocrit
Time until impaired plasma refill rate | 48 h
blood pressure | Changes from Baseline to 48 h after intervention
heart rate | Changes from Baseline to 48 h after intervention
Serum Creatinine level | 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Westenfeld, MD, Principal Investigator — Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Dusseldorf; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Dusseldorf
Locations (1):
- Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Dusseldorf, Düsseldorf, Germany